CLINICAL TRIAL: NCT03249688
Title: Multimodal Preventive Trial for Alzheimer's Disease (MIND-ADmini Pilot Trial)
Brief Title: Multimodal Preventive Trial for Alzheimer's Disease
Acronym: MIND-ADmini
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Eastern Finland (Other); Universität des Saarlandes (Other); University Hospital, Toulouse (Other)
Responsible Party: Principal Investigator, Miia Kivipelto, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E0750301
Record Dates: First submitted 2017-07-08; First posted 2017-08-15 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Alzheimer Disease; Prodromal
Keywords: Lifestyle intervention; Medical food; Randomized controlled trial; Prodromal Alzheimer's disease; Prevention; Intervention; Multidomain; Multimodal
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): Regular health advice
  Interventions: Other: Regular health advice
- Multidomain 1 (Experimental): Multidomain lifestyle
  Interventions: Behavioral: Multidomain lifestyle
- Multidomain 2 (Experimental): Multidomain lifestyle + medical food
  Interventions: Behavioral: Multidomain lifestyle; Dietary Supplement: Medical food

INTERVENTIONS:
Other: Regular health advice — Routine healthy lifestyle counseling
  Arms: Control
Behavioral: Multidomain lifestyle — Nutritional guidance, exercise, cognitive training, vascular risk monitoring
  Arms: Multidomain 1; Multidomain 2
Dietary Supplement: Medical food — Medical food product (Fortasyn Connect)
  Arms: Multidomain 2

SUMMARY:
The main aim of the MIND-ADmini pilot trial is to evaluate the feasibility of a multimodal lifestyle intervention among patients with prodromal AD.

DETAILED DESCRIPTION:
Given the multifactorial etiology of Alzheimer's disease (AD), multimodal interventions targeting several risk factors and disease mechanisms simultaneously are most likely to be effective for preventing dementia. Multimodal lifestyle interventions have so far been tested in at-risk older adults from the general population, but not in patients with prodromal AD.

The main aim of the MIND-ADmini pilot trial is to evaluate the feasibility of a multimodal lifestyle intervention among individuals with prodromal AD.

This 6-month pilot trial is planned to include 150 participants randomized into 3 arms:

1. Control (regular health advice)
2. Multidomain lifestyle intervention (nutritional guidance, exercise, cognitive training and monitoring and management of vascular and metabolic risk factors)
3. Multidomain lifestyle intervention + medical food. The multidomain lifestyle intervention is adapted from the Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER, NCT01041989). The medical food product includes the specific multi-nutrient combination Fortasyn Connect (containing the omega-3 fatty acids docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA), uridine monophosphate, choline, vitamins B12, B6, C, E, and folic acid, phospholipids, and selenium). The rationale for combining a multidomain lifestyle intervention with medical food is evidence indicating synergistic effects between different intervention components (e.g. omega-3 fatty acids and physical activity). Nutrient deficiencies have been described in AD, and medical food may be needed in addition to dietary guidance for optimal effect. The use of Fortasyn Connect alone in prodromal AD has been investigated in another clinical trial (www.lipididiet.eu), and thus this arm is not included in MIND-ADmini.

The 6-month MIND-ADmini pilot trial will be conducted in Sweden, Finland, Germany and France. An additional 6-month optional extension of the pilot trial will also be considered.

Primary outcome is feasibility of the multimodal intervention. Secondary outcomes include adherence to intervention components (intervention arms), and adherence to healthy lifestyle changes (all arms). Detailed cognitive assessments (Neuropsychological Test Battery, NTB) and functional assessments (Clinical Dementia Rating, CDR; and Alzheimer's Disease Cooperative Study-Activities of Daily Living, ADCS-ADL) will also be conducted at baseline and 6-month visit for the purpose of obtaining reliable estimates of change over time for power calculations for a future larger multimodal intervention trial (MIND-ADmaxi).

ELIGIBILITY:
Inclusion criteria:

A) Prodromal AD as defined as -1 SD on 2 out of 8 tests, at least 1 memory:

Memory FCSRT - delayed free recall* ≤ 8 FCSRT free recall - learning ≤ 22 WMS-R story delayed recall (%) ≤75% WMS-R delayed recall of figures (%) ≤ 75% *Free and Cued Selective reminding test

Non-memory TMT A ≥ 60 TMT B ≥ 150 Symbol Digit Substitution Test ≤ 35 (120 sec.) Category Fluency ≤ 16 (60 sec.)

* Evidence for underlying AD pathology within 2 year prior to screening by either:

  1. CSF beta amyloid 1-42/1-40x10 ratio<1 and/or elevated T-tau and/or elevated phospho-tau and/or low beta amyloid 42 based on local lab cut-offs OR
  2. MRI evidence for medial temporal lobe atrophy (MTA score 1 or higher) OR
  3. Abnormal FDG PET and/or PiB PET compatible with AD type change

     B) Potential for lifestyle improvement, defined according to a Lifestyle Index.

     Lifestyle index. Participants with a score of 3 or above are included in the study.

     The lifestyle index identifies individuals who do not already have very healthy lifestyles, and thus have a margin for improving their lifestyle based on the MIND-AD intervention. The score is calculated by adding 1 point for each of the following factors:
* Physical activity less than 2.5 hours a week (defined as physical activity intensive enough to lead to sweating and some breathlessness)
* Diet - less than 5 portions of fruits and vegetables per day
* Diet - less than 2 portions of fish per week
* Hypertension (diagnosed by physician or current antihypertensive treatment or
* SBP>140mmHg or DBP>90 mmHg)
* Diabetes (type 1 or 2 diagnosed by physician; or current diabetes medication; or recorded elevated fasting blood glucose or HbA1C as per local guidelines within the past 6 months)
* Ongoing symptoms of sleep problems, depressive symptoms or psychological stress symptoms for at least 1 month, judged by the clinician as having some impact on everyday life

C) Age 60-85 D) MMSE ≥ 24 E) Availability of a responsible study partner. F) Written informed consent from participant as well as study partner G) Putative prescription cognitive enhancers (e.g. ginkgo, cholinesterase inhibitors) and statins are not excluded but the dosage should be stable prior to randomization. Doses should be kept stable during the study if possible.

Exclusion criteria

* Dementia according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* Use of omega-3 preparations > 500mg EPA+DHA per day
* Alcohol or drug abuse
* A concomitant serious disease
* Major depressive disorder (DSM-IV)
* Regular intake of supplements for vitamin B6, B12, folic acid, vitamin C and/or E > 200% RDI, unless prescribed by physician
* Participation in any other clinical trial in the last 30 days
* Subjects with MRI (or CT) scan consistent with a diagnosis of stroke, intracranial bleeding, mass lesion or NPH. Those subjects with a MRI scan demonstrating minimal white matter changes (Fazekas scale for white matter lesions <=3) and up to 1-2 lacunar infarcts which are judged to be clinically insignificant are allowed
* Severe loss of vision or communicative ability
* Conditions preventing cooperation as judged by the study physician
* Concomitant participation in any intervention trial

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  Recruitment rate of participants within a 6 months period
Overall adherence to the intervention | 6 months
  Overall adherence to the intervention during 6 months
Retention rate | 6 months
  Retention rate of participants during 6 months

SECONDARY OUTCOMES:
Adherence to intervention components | 6 months
  Intervention arms only
Adherence to healthy lifestyle changes | 6 months
  All arms

OTHER OUTCOMES:
Change in Body Mass Index | 6 months
  Height (cm) and weight (kg) are used to calculate Body Mass Index
Change in Hip-waist ratio | 6 months
  Hip and waist measurements (cm) are used for hip-waist ratio calculations
Change in blood pressure | 6 months
  Including measurements of systolic blood pressure, diastolic blood pressure, and pulse pressure
Change in blood lipids | 6 months
  Including measurements of serum total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides
Change in glucose metabolism markers | 6 months
  Including measures of glucose, insulin, HbA1c
Change in inflammation | 6 months
  CRP measures
Depressive symptoms | 6 months
  Geriatric Depression Scale
Stress-related symptoms | 6 months
  Perceived Stress Scale
Physical performance | 6 months
  Timed 10-meter dual-task test & Short Physical Performance Battery (SPPB)
Health-related quality of life | 6 months
  RAND36
Blood biomarkers | 6 months
  e.g lipid metabolism, inflammation, vitamins (e.g D & B)
Self-reported adherence to each intervention component | 6 months
  The following intervention components: nutrition, exercise, cognitive training, monitoring of vascular factors

CONTACTS AND LOCATIONS:
Overall Officials: Miia Kivipelto, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Cummings J, Scheltens P, McKeith I, Blesa R, Harrison JE, Bertolucci PH, Rockwood K, Wilkinson D, Wijker W, Bennett DA, Shah RC. Effect Size Analyses of Souvenaid in Patients with Alzheimer's Disease. J Alzheimers Dis. 2017;55(3):1131-1139. doi: 10.3233/JAD-160745. PMID 27767993
- [Background] Dubois B, Feldman HH, Jacova C, Dekosky ST, Barberger-Gateau P, Cummings J, Delacourte A, Galasko D, Gauthier S, Jicha G, Meguro K, O'brien J, Pasquier F, Robert P, Rossor M, Salloway S, Stern Y, Visser PJ, Scheltens P. Research criteria for the diagnosis of Alzheimer's disease: revising the NINCDS-ADRDA criteria. Lancet Neurol. 2007 Aug;6(8):734-46. doi: 10.1016/S1474-4422(07)70178-3. PMID 17616482
- [Background] van Wijk N, Broersen LM, de Wilde MC, Hageman RJ, Groenendijk M, Sijben JW, Kamphuis PJ. Targeting synaptic dysfunction in Alzheimer's disease by administering a specific nutrient combination. J Alzheimers Dis. 2014;38(3):459-79. doi: 10.3233/JAD-130998. PMID 23985420
- [Derived] Levak N, Lehtisalo J, Thunborg C, Westman E, Andersen P, Andrieu S, Broersen LM, Coley N, Hartmann T, Irving GF, Mangialasche F, Ngandu T, Pantel J, Rosenberg A, Sindi S, Soininen H, Solomon A, Wang R, Kivipelto M. Nutrition guidance within a multimodal intervention improves diet quality in prodromal Alzheimer's disease: Multimodal Preventive Trial for Alzheimer's Disease (MIND-ADmini). Alzheimers Res Ther. 2024 Jul 3;16(1):147. doi: 10.1186/s13195-024-01522-8. PMID 38961421
- [Derived] Thunborg C, Wang R, Rosenberg A, Sindi S, Andersen P, Andrieu S, Broersen LM, Coley N, Couderc C, Duval CZ, Faxen-Irving G, Hagman G, Hallikainen M, Hakansson K, Kekkonen E, Lehtisalo J, Levak N, Mangialasche F, Pantel J, Rydstrom A, Stigsdotter-Neely A, Wimo A, Ngandu T, Soininen H, Hartmann T, Solomon A, Kivipelto M. Integrating a multimodal lifestyle intervention with medical food in prodromal Alzheimer's disease: the MIND-ADmini randomized controlled trial. Alzheimers Res Ther. 2024 May 30;16(1):118. doi: 10.1186/s13195-024-01468-x. PMID 38812047